CLINICAL TRIAL: NCT05483712
Title: A Clinical Trial to Assess Skin Dose in Post-mastectomy Adjuvant Radiation Therapy of Breast Cancer Patients Using a Brass Mesh Bolus
Brief Title: Brass Mesh Bolus in Rotational Post-Mastectomy Radiation Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Cancer Centre (Other)
Collaborators: Hannah Dahn (Unknown)
Responsible Party: Principal Investigator, Thalat Monajemi, Medical Physicist, Nova Scotia Cancer Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12341234
Record Dates: First submitted 2022-07-25; First posted 2022-08-02 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Radiation Therapy; Brass Mesh; Bolus; Skin Dose
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a single-site study designed to generate data quantifying the skin dose under brass mesh bolus.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Post-Mastectomy Radiation Therapy Patients (Experimental): Any patient who is going through radiation to their chest wall following mastectomy using a rotational delivery technique and 6 MV, and uses Superflab bolus for some but not all fractions of radiotherapy
  Interventions: Device: Brass Mesh Bolus

INTERVENTIONS:
Device: Brass Mesh Bolus — During a standard-of-care 15 fraction radiotherapy treatment, a brass mesh bolus will be used for a single fraction. Small in-vivo dosimeters will be used for three treatment fractions to measure and compare skin doses for quantification purposes.

SUMMARY:
The hypothesis is that the daily use of brass mesh bolus achieves a comparable dose to every-other-day use of Superflab bolus (current standard of care) in chest wall post-mastectomy patients treated with rotational 6 MV photon delivery.

DETAILED DESCRIPTION:
Intervention: During a standard-of-care 15 fraction radiotherapy treatment, a brass mesh bolus will be used for a single fraction. Small in-vivo dosimeters will be used for three treatment fractions to measure and compare skin doses for quantification purposes.

Comparator: Superflab and no bolus applied as per the treating physician's practice, typically on alternate days. The intervention and comparator tools are to be utilized on each participant.

Primary outcome

1. To determine the skin dose under brass mesh bolus and compare it with the skin dose under Superflab bolus (current standard of care).
2. To determine the number of fractions for which brass mesh bolus should be used to achieve an acceptable skin dose.

ELIGIBILITY:
Inclusion Criteria:

Women undergoing rotational chest wall radiotherapy following mastectomy for breast cancer treatment who would utilize Superflab bolus on some, but not all, days of radiotherapy treatment.

Exclusion Criteria:

Patients who require daily bolus due to skin involvement or other high-risk features requiring a high skin dose will not be included.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-11-21 (Estimated); Study Completion 2024-11-21 (Estimated)

PRIMARY OUTCOMES:
Skin Dose Enhancement Under Brass Mesh Bolus | through study completion, an average of 1 year
  During days one, two, and three of radiation therapy, patients on this study utilize no-bolus, 5-mm thick Superflab bolus, and brass mesh bolus, respectively. Each day, nine in-vivo dosimeters (OSLDs) will be placed on patient skin to sample the skin dose in cGy. As a result, for each patient on this study, skin dose enhancement of brass mesh compared with no-bolus can be related to that of Superflab bolus. At the end of the study, the average and range of skin dose enhancement under brass mesh bolus for a sample size of twenty patients will be reported.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada

IPD SHARING:
Plan to Share IPD: Yes